CLINICAL TRIAL: NCT01869413
Title: Tranexamic Acid During Cystectomy Trial (TACT)
Acronym: TACT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Dalhousie University (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Laval University (Other); University of Western Ontario, Canada (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIHR MOP-342559; Control # 162042 (Other: Health Canada)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Bladder Cancer
Keywords: urothelial cell carcinoma; transition cell carcinoma; bladder cancer; radical cystectomy; cystectomy; bladder removal; tranexamic acid; cyklokapron
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Tranexamic acid will be administered as an intravenous infusion of 10 mg/kg over 10 minutes (loading dose) prior to surgical incision, followed by 5 mg/kg/hour continuous maintenance infusion for the length of surgery (typically 4 to 8 hours). For example, an 80 kg patient would receive 800 mg prior to incision and a 400 mg/hr infusion for the duration of surgery. For a 6 hour procedure, the total dose administered would be 3200 mg.
  Interventions: Drug: Tranexamic Acid
- Placebo control (Placebo Comparator): As there is no standard of care concerning administration of anti-fibrinolytic agents in cystectomy procedures, controls will follow the same dosing and schedule as above (loading dose followed by maintenance infusion), but with 0.9% sodium chloride.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid will be administered as an intravenous infusion of 10 mg/kg over 10 minutes (loading dose) prior to surgical incision, followed by 5 mg/kg/hour continuous maintenance infusion for the length of surgery (typically 4 to 8 hours).
  Other Names: Cyklokapron (Pfizer)
  Arms: Tranexamic Acid
Drug: Placebo — As there is no standard of care concerning administration of anti-fibrinolytic agents in cystectomy procedures, controls will follow the same dosing and schedule as above (loading dose followed by maintenance infusion), but with 0.9% sodium chloride.
  Other Names: Normal Saline
  Arms: Placebo control

SUMMARY:
A cystectomy is the removal of the bladder and adjacent organs in patients with bladder cancer. This often results in significant blood loss, and about 60% of patients will require a blood transfusion during or up to 30 days after surgery. Significant blood loss may result in cardiovascular morbidity, and the use of blood products are expensive and expose patients to risk.

Tranexamic acid reduces breakdown of hemostatic blood clots and it has therapeutic benefit when used in other surgical procedures to reduce blood loss and the need for transfusion. The current study will be the first to evaluate whether tranexamic acid is effective and safe to use during radical cystectomy. The results of the study will have an immediate impact on patient care.

DETAILED DESCRIPTION:
Removal of the bladder and adjacent organs in patients with bladder cancer (radical cystectomy) often results in significant blood loss, and approximately 60% of patients require peri-operative blood transfusion. Reducing blood loss and the frequency of transfusion offers several benefits, including donor blood conservation, health care cost reduction, and avoidance of blood product exposure. Tranexamic acid is an amino acid lysine derivative with strong antifibrinolytic clotting properties that can be administered systemically. This medication has been used in a variety of operative procedures, notably in high risk cardiac surgery, to decrease peri-operative blood loss, and it is associated with an acceptable risk of adverse events. Systemic anti-hemorrhagics are infrequently used during radical cystectomy, and to the investigators knowledge their effects have not been evaluated in a clinical trial.

Overall objective: To conduct a randomized controlled trial of systemic tranexamic acid compared to placebo in reducing the number of blood transfusions in patients undergoing radical cystectomy for bladder cancer.

Design: A multi-center, randomized, double-blinded, placebo controlled trial.

Study population: Consenting patients 18 years of age and older undergoing a radical cystectomy for bladder cancer, excluding those who: are unwilling to receive blood products due to personal reasons, are pregnant, have active angina, have a known allergy to tranexamic acid, or have a known personal history of deep venous thrombosis, atrial fibrillation, coronary stent, sub-arachnoid hemorrhage, pulmonary embolism, thrombotic stroke and / or acquired disturbance of colour vision. The study will recruit 354 patients from Dalhousie University, McGill University, Université de Montreal, Université Laval, University of Ottawa, University of Western Ontario and University of Alberta.

Intervention:

Tranexamic Acid arm: Tranexamic acid will be administered as an intravenous infusion of 10 mg/kg within 10 minutes (loading dose) and before surgical incision, followed by 5 mg/kg/hour continuous maintenance infusion for the length of surgery (typically 4 to 8 hours). For example, an 80 kg patient would receive 800 mg prior to incision and a 400 mg/hour infusion for the duration of surgery. For a 6 hour procedure, the total dose administered would be 3200 mg.

Placebo arm: As there is no standard of care concerning administration of antifibrinolytic agents in cystectomy procedures, controls will follow the same dosing and schedule described above, but with 0.9% saline infusion.

Outcomes: The primary research objective is whether the use of systemic tranexamic acid compared to placebo reduces the proportion of radical cystectomy patients requiring red blood cell transfusion up to 30 days post-operative (from a 50% transfusion rate with placebo to 35% with tranexamic acid). Secondary questions are: Will use of systemic tranexamic acid compared to placebo result in reductions in: i) intraoperative blood loss, ii) amounts of transfused blood products, and iii) post-operative complications? The safety (thrombotic events) of tranexamic acid will also be evaluated.

Importance of this study: If tranexamic acid reduces the number of blood transfusions, there will be an immediate impact to cystectomy patients, and surgeons may consider the routine use of systemic tranexamic acid during similar abdomino-pelvic procedures associated with significant blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Participant ≥ 18 years at time of consent
* Participant has bladder cancer and will undergo radical cystectomy to remove bladder
* Participant is willing to receive blood products (i.e. packed red blood cells, platelets, plasma)
* Have obtained Informed Consent

Exclusion Criteria:

* Participant declines consent
* Participants incapable (incompetent) of providing Informed Consent
* Participant is under 18 years
* Participant is unwilling to receive blood products due to personal reasons
* Participant has thromboembolic disease (active or diagnosed within 1 year) such as deep vein thrombosis, pulmonary embolism or cerebral thrombosis)
* Participant with known personal history of subarachnoid haemorrhage.
* Participant has acquired disturbances to his / her colour vision (does not apply to congenital colour blindness)
* Participant is pregnant (confirmed by βHCG test)
* Participant has a known allergy to tranexamic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2013-06; Primary Completion 2021-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients transfused at least one unit of packed red blood cell transfusion | up to 30 days post-operative

SECONDARY OUTCOMES:
total units of red blood cells transfused | up to 30 days post-operative
occurrence of postoperative bleeding requiring intervention | up to 30 days post-operative
  intervention noted as reoperation or angioinfarction
occurrence of platelet transfusion | up to 30 days post-operative
total units of platelets transfused | up to 30 days post-operative
occurrence of plasma transfusion | up to 30 days post-operative
total units of plasma transfused | up to 30 days post-operative
estimated intra-operative blood loss | up to 30 days post-operative
change in hemoglobin | up to 30 days post-operative

OTHER OUTCOMES:
occurrence of severe adverse events | up to 30 days post-operative
number of treatment failures | up to 30 days post-operative
  treatment failures noted as the need for anti-hemorrhagic rescue interventions such as topical agents (oxidized cellulose) and recombinant Factor VIIa

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Breau, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (10):
- Canada (10):
  - Northern Alberta Urology Centre, Edmonton, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Complex (LHSC), London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Centre Hospitalier de l'Université de Québec (CHUQ), Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breau RH, Lavallee LT, Cagiannos I, Momoli F, Bryson GL, Kanji S, Morash C, Turgeon AF, Zarychanski R, Houston BL, McIsaac DI, Mallick R, Knoll GA, Kulkarni G, Izawa J, Saad F, Kassouf W, Fradet V, Rendon R, Shayegan B, Fairey A, Drachenberg DE, Fergusson D. Tranexamic Acid During Radical Cystectomy: A Randomized Clinical Trial. JAMA Surg. 2024 Dec 1;159(12):1355-1363. doi: 10.1001/jamasurg.2024.4183. PMID 39356537
- [Derived] Breau RH, Lavallee LT, Cnossen S, Witiuk K, Cagiannos I, Momoli F, Bryson G, Kanji S, Morash C, Turgeon A, Zarychanski R, Mallick R, Knoll G, Fergusson DA. Tranexamic Acid versus Placebo to Prevent Blood Transfusion during Radical Cystectomy for Bladder Cancer (TACT): Study Protocol for a Randomized Controlled Trial. Trials. 2018 May 2;19(1):261. doi: 10.1186/s13063-018-2626-3. PMID 29716640
- See also: Tranexamic Acid (Cyklokapron) Product Monograph — https://www.pfizer.ca/cyklokapron-tranexamic-acid